CLINICAL TRIAL: NCT05729412
Title: A Prescription Audit In The Outpatient Department Of Nabh & Jci Approved Super Speciality Hospital In The Capital Territory Of India
Brief Title: Prescription Audit in OPD of NABH & JCI Approved Hospital in Capital Territory of India
Status: Completed | Type: Observational
Sponsor: Kakatiya University (Other)
Responsible Party: Principal Investigator, Satyam Suman, Clinical Pharmacy Department, Kakatiya University
Other Study IDs: MAX/IEC/2022/NOV/PA01
Record Dates: First submitted 2023-01-31; First posted 2023-02-15 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Quality of Life
Keywords: Medical Audit; Prescription Audit; Gender difference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Compliance: Prescription is filled for specific parameters
  Interventions: Other: Mentioned
- Non-compliance: Prescription is not filled for specific parameters
  Interventions: Other: Mentioned
- Not available - NA: Data not available
  Interventions: Other: Mentioned

INTERVENTIONS:
Other: Mentioned — If prescription is properly filled for specific details than it is compliance
  Other Names: Prescription is properly filled

SUMMARY:
Aim of the study: The aim of the study is to evaluate the quality of the prescription provided to the outpatient.

Need of study:

For the promotion of the good clinical practice To improve the efficiency of the multidisciplinary team in the healthcare To utilize resources to provide better patient care To improve quality standards and quality of care For implication of professional practices To identify and eliminate deficient practice

Objectives:

1. To study the quality of good prescription
2. In minimization of prescription errors and medication errors
3. Also to comply with good clinical practice
4. Enhancement of patient safety
5. In the maintenance of rational prescribing
6. To study the quality of care provided by the hospital to the patient

Plan of study:

* To select the patient based on inclusion and exclusion criteria
* To collect the information from OP's prescription
* To identify prescribing errors and medication error
* To study the management of good prescription

Study Sites: Max Super Speciality Hospital, Saket, New Delhi (INDIA) Study Design: Observational cohort study Study Duration: 1 month (November 2022)

DETAILED DESCRIPTION:
Source of the data: Review of out-patient prescription Sample size: 100 prescription

Possible outcomes:

Minimization of prescribing errors It improves the quality of care Enhancement of patient safety Compliance with good clinical practice In the maintenance of rational prescribing

ELIGIBILITY:
Inclusion Criteria:

* Participants who are willing to participate.
* Participants who are attending in the out-patient department.
* Participants reported during the study period.
* Participants who have a prescription which is legible and complete.

Exclusion Criteria:

* Participants who are unwilling to provide the required information.
* Participants who are not attending the out-patient department.
* Participants whose prescription is not legible and competent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient prescription which is randomly picked during study period
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Percentage of prescription | November 01, 2022 to November 30, 2022
  Data is available sufficient

CONTACTS AND LOCATIONS:
Locations (1):
- Max Super Speciality Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
If planned, definitely it would be notified